CLINICAL TRIAL: NCT04217655
Title: Low-dose Computed Tomography-guided Core Needle Biopsy for Lung Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20200102-001
Record Dates: First submitted 2020-01-01; First posted 2020-01-03 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Lung Cancer; Lung; Node
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose computed tomography group (Experimental): Patients undergo low-dose computed tomography-guided lung biopsy for lung nodule on day 1.
  Interventions: Diagnostic Test: Low-dose computed tomography
- Standard-dose computed tomography group (Active Comparator): Patients undergo standard-dose computed tomography-guided lung biopsy for lung nodule on day 1.
  Interventions: Diagnostic Test: Standard-dose computed tomography

INTERVENTIONS:
Diagnostic Test: Low-dose computed tomography — Radiation dose under the low-dose protocol computed tomography (120 kilovolt, 15 milliampere seconds)
  Arms: Low-dose computed tomography group
Diagnostic Test: Standard-dose computed tomography — Radiation dose under the standard-dose protocol computed tomography (120 kilovolt, 150 milliampere seconds)
  Arms: Standard-dose computed tomography group

SUMMARY:
Investigators aim to compare the diagnostic accuracy and radiation exposure between low-dose and standard-dose computed tomography-guided core needle biopsy for lung nodules.

DETAILED DESCRIPTION:
At present, low-dose scanning protocol is widely used in computed tomography-guided interventions because these procedures usually require repeat scans, which causes more radiation exposure to the patients. Computed tomography-guided core needle biopsy is widely used in diagnosis of lung nodules with an overall diagnostic accuracy of 93%-97%. Compared with the large lung lesions, computed tomography-guided core needle biopsy for lung nodules might require more scanning to adjust the position of needle tip. Therefore, it might expose the patients to more radiation. However, studies regarding computed tomography-guided core needle biopsy for lung nodules are still lacking.

In this study, investigators aim to compare the diagnostic accuracy and radiation exposure between low-dose and standard-dose computed tomography-guided core needle biopsy for lung nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Non-diagnostic lung lesions (no definitive pathological diagnosis);
2. Lesion size between 5 and 30 mm;
3. Solid lung lesions.

Exclusion Criteria:

1. The lesion which has been punctured previously;
2. A lesion that had shrunk in size or a lesion with a stable size for 1 year;
3. Severe dysfunction in heart, lung and coagulation function;
4. Patients who refused to provide informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | From the date of randomization until the date of first documented final diagnosis, assessed up to 12 months
  Diagnostic accuracy is defined as the biopsy diagnosis matches with the final diagnosis. The final diagnosis is made according to the surgical or follow-up findings.

SECONDARY OUTCOMES:
Radiation dose | From the date of randomization until the date of first documented biopsy procedures, assessed up to 1 day.
  Radiation dose is the radiation exposure from the computed tomography device to patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Chi Li, MD, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Fu YF, Li GC, Xu QS, Shi YB, Wang C, Wang T. Computed tomography-guided lung biopsy: a randomized controlled trial of low-dose versus standard-dose protocol. Eur Radiol. 2020 Mar;30(3):1584-1592. doi: 10.1007/s00330-019-06464-6. Epub 2019 Nov 27. PMID 31776740
- [Derived] Li EL, Ma AL, Wang T, Fu YF, Liu HY, Li GC. Low-dose versus standard-dose computed tomography-guided biopsy for pulmonary nodules: a randomized controlled trial. J Cardiothorac Surg. 2023 Mar 16;18(1):86. doi: 10.1186/s13019-023-02183-8. PMID 36927419